CLINICAL TRIAL: NCT05803603
Title: Social Work Assistance and Stipends for Housing (SASH): Improving Outcomes for Homeless Patients Receiving Methadone for Opioid Use Disorder
Brief Title: Social Work Assistance and Stipends for Housing (SASH)
Acronym: SASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, George Unick, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00100771
Record Dates: First submitted 2023-03-23; First posted 2023-04-07 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Opioid-Related Disorders; Housing Problems
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: 8 individuals will be recruited and followed for 12 months following the intervention. The intervention includes providing a $500 monthly housing stipend for six months and twelve months of social work support to find permanent housing. Individuals will be asked to provide information thought interviews and clinical records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Individuals will receive $500 monthly stipend for the first months of the study and will receive twelve months of social work supports to help individuals find permanent housing.
  Interventions: Behavioral: Stipend and Social Work Supports

INTERVENTIONS:
Behavioral: Stipend and Social Work Supports — Same as arm description

SUMMARY:
SASH is a clinical trial feasibility study that will provide an intervention to improve Opioid Use Disorder (OUD), Quality of Life (QOL), and housing outcomes for homeless patients receiving Medication for Opiate Use Disorder (MOUD). The main questions of the study are does a $500 housing stipend for individuals on MOUD increase treatment retention, improved quality of life and prevent homelessness.

DETAILED DESCRIPTION:
SASH is a clinical trial feasibility study that will provide an housing stipend for 8 individuals (N=8) experience homelessness and currently being treated for OUD to improve OUD treatment outcomes, QOL, and housing outcomes. To achieve these goals, patients will receive monthly $500 housing stipends that can be used for a broad range of temporary housing included in a list of resources compiled by the study. These stipends will be accompanied by Social Work assistance to find permanent housing which will last the full 12 months of the study. SASH will recruit OUD patients receiving MOUD who are struggling with homelessness, defined as living in an emergency shelter or a place not meant for habitation instead of a fixed, regular, and adequate nighttime residence. This definition is consistent with the one used by the U.S. Department of Housing and Urban Development. The patients will be recruited from the University of Maryland Addiction Treatment Program (ATP), a certified Substance Use Disorder (SUD) treatment program that provides MOUD and collocates medical care, wellness programs, and research. Patients will be eligible for SASH if they experienced homelessness during at least 15 of the 30 days preceding the dispensing of the first month's stipends.SASH will accomplish its goals using the following aims and objectives:

AIM 1: Improve OUD outcomes

* Hypothesis 1a: Patients will miss fewer methadone doses and receive more take-home methadone doses after receiving the stipends and Social Work assistance Endpoint: Percentages of missed and take-home methadone doses, as recorded by the software tracking methadone-dispensing at the ATP, in the 3-month period before the study, between Month 3 and 6 of the study, and between Month 9 and 12 of the study
* Hypothesis 1b: Patients will experience an improvement in their OUD after receiving the stipends and Social Work assistance Endpoint: OUD Checklist scores completed at Day 0, Month 6, and Month 12 of the study
* Hypothesis 1c: Patients will use fewer opioids and illicit substances after receiving the stipends and Social Work assistance Endpoint: Monthly urine toxicology tests (UTT) three months before study entry and monthly during the study

AIM 2: Improve QOL

* Hypothesis 2a: Patients will experience improvement in QOL during the study Endpoint: SF-36 scores at Day 0, Month 6, and Month 12 of the study
* Hypothesis 2b: Patients will report benefit from receiving the stipends and Social Work assistance

AIM 3: Prevent homelessness

* Hypothesis 3a: The monthly $500 stipends will prevent patients from being homeless Endpoint: Percentage of days patients are homeless during the 6-month period stipends are distributed
* Hypothesis 3b: Patients will be in housing by the end of the study Endpoint: Percentage of patients who are homeless or in either permanent or temporary housing by Month 12 of the study

ELIGIBILITY:
Inclusion Criteria:

* Experienced homelessness during at least 15 of the 30 days preceding enrollment
* Is a patient at the University of Maryland Addiction Treatment Program (ATP) receiving methadone treatment.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Addiction Treatment Program (ATP), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made available to other researchers. Because only a small number of participants are being enrolled (N=8) outcomes data will be limited to what can be share without identifying individuals.
Supporting Information: Study Protocol
Time Frame: The data will be available at the end of the study period for 5 years.
Access Criteria: Access criteria to be determined.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 8
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean of Age
  years | 46.75 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Methadone Doses
Description: Percentage of Missed Methadone Doses, Range 0 - 100%, Lower percentages mean better outcome.
Time Frame: 3 months prior to enrollment
Measure: Mean (Standard Deviation); unit: percent of missed doses
Arm/Group | Intervention Arm
Number analyzed (Participants) | 8
percent of missed doses | 4.58 (4.58)

2. Primary Outcome: Methadone Doses
Description: Percentage of Missed Methadone Doses, Range 0 - 100%, Lower percentages mean better outcome.
Time Frame: 3-6 months post enrollment
Measure: Mean (Standard Deviation); unit: Percent Missed
Arm/Group | Intervention Arm
Number analyzed (Participants) | 7
Percent Missed | 7.47 (7.94)

3. Primary Outcome: Methadone Doses
Description: Percentage of Missed Methadone Doses, Range 0 - 100%, Lower percentages mean better outcome.
Time Frame: 9-12 months post enrollment.
Measure: Mean (Standard Deviation); unit: Percent Missed
Arm/Group | Intervention Arm
Number analyzed (Participants) | 7
Percent Missed | 34.11 (32.11)

4. Primary Outcome: OUD Checklist Scores
Description: Scores on the Diagnostic and Statistical Manual V OUD checklist. Range 0 - 13. Higher scores mean worse outcome with 2-3 as mild severity, 4-5 moderate severity and 6 or more as severe.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 8
units on a scale | 8.25 (7.4)

5. Primary Outcome: OUD Checklist Scores
Description: as for outcome 4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
units on a scale | 7.4 (4.4)

6. Primary Outcome: OUD Checklist Scores
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
units on a scale | 7.2 (5.3)

7. Primary Outcome: Urine Toxicology Tests
Description: Detection of positive urine toxicology tests collected from chart reviews. Values are positive or negative for controlled substances. Positive test the worse outcome
Time Frame: Three months prior to enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 8
Participants | 7

8. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 7
Participants | 5

9. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 4

10. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 5

11. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 5

12. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 7
Participants | 6

13. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 6

14. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 5

15. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 8
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 5

16. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 9
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 6

17. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 10
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 5

18. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 11
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
Participants | 3

19. Primary Outcome: Urine Toxicology Tests
Description: as for outcome 7
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 4
Participants | 3

20. Primary Outcome: Quality of Life Scores
Description: SF-36 scores 0 (worst) to 100 (best)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 8
units on a scale | 34.4 (14.5)

21. Primary Outcome: Quality of Life Scores
Description: SF-36 scores 0 (worst) to 100 (best)
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
units on a scale | 31 (10.8)

22. Primary Outcome: Quality of Life Scores
Description: SF-36 scores 0 (worst) to 100 (best)
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
units on a scale | 32 (10.4)

23. Primary Outcome: Housed vs Unhoused at 6 Months
Description: Count of participants that are housed at 6 months
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 6
Participants | 4

24. Primary Outcome: Housed vs Unhoused at 6 Months
Description: Count of housed at 12 month
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
Participants | 3
Statistical Analysis 1: Comparison: Intervention Arm; We recruited 8 homeless individuals and followed them for 12 months. 4 individuals (50%) were housed at 6 months and 3 (37.5) were housed at 12 months; Test type: Superiority; p = .125, McNemar; Odds Ratio (OR) = 2.0, 95% CI 2-sided [.37 to 10.92]; See results above

ADVERSE EVENTS:
Time Frame: Data were collected for 12 months.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05803603/Prot_SAP_000.pdf